CLINICAL TRIAL: NCT05745532
Title: Safety and Efficacy Evaluation of β-globin Restored Autologous Hematopoietic Stem Cells in β-thalassemia Major Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shenzhen Hemogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SZ-101; NCT04592458 (obsolete NCT alias)
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: β-thalassemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Ten transfusion-dependent β-thalassaemia subjects aged 8-16 years will be reinfused with β-globin-restored autologous hematopoietic stem cells modified with LentiHBBT87Q.
  Interventions: Biological: β-globin restored autologous hematopoietic stem cells

INTERVENTIONS:
Biological: β-globin restored autologous hematopoietic stem cells — β-globin-restored autologous hematopoietic stem cells modified with LentiHBBT87Q

SUMMARY:
This is an open label study to evaluate the safety and efficacy of β-globin Restored Autologous Hematopoietic Stem Cells in ß-Thalassemia Major Patients

DETAILED DESCRIPTION:
We will recruit ß-thalassaemia major patients and collect their autologous hematopoietic stem cells, which will be modified with the LentiHBBT87Q system to restore β-globin expression. After conditioning, the autologous hematopoietic stem cells with restored β-globin will be reinfused to the patients and followed up for two years to collect data.

ELIGIBILITY:
Inclusion Criteria:

* 8-16 years old. Subject and/or subject's legal guardian fully understand and voluntarily sign informed consent;
* Clinically diagnosed as transfusion-dependent β-thalassemia major;
* With sufficient RBC infusion, subjects must maintain hemoglobin ≥9g/dL, serum ferritin threshold ≤ 3000 ng/mL and the liver iron overload mild or absent for at least 3 months before mobilization of hematopoietic stem cell;
* Follow the arrangements for treatment and regular medical checks within two years post-transplantation

Exclusion Criteria:

* The physical condition does not meet the requirements for hematopoietic stem cell mobilization and transplantation myeloablation;
* Received gene therapy and allogeneic HSCT in the past.
* Have an available HLA matched donor.
* Enrolling in another clinical trial.
* Other unsuitable conditions identified by doctors.

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Frequency and severity of adverse events (AEs) and serious adverse events (SAEs) | 0-100 days
  The number and the percentage of adverse events related to transplantation in 100 days will be summarized according to NCI CTCAE 5.0
Overall survival | 0-24 months
  Number of patients alive through the whole trial will be record
Proportion of engraftment | 0-24 months
  Neutrophil count [ANC] >=500 /mm3 for 3 consecutive days and platelet count [PLT] >20,000/mm3 for7 consecutive days
Replication competent lentivirus (RCL) | 0-24 months
  The percentage of RCL should be negative in the 24 months after transplant
Dynamics of viral integration sites (VIS) | 0-24 months
  Evaluation of the percentage of participants without abnormal clonal proliferation and polyclonal engraftment . More than 1000 VIS retrieved from peripheral blood should be checked.

SECONDARY OUTCOMES:
The average Insertion copy number (VCN) in peripheral blood mononuclear cells | 18-24 Months
  The average insertion copy number (VCN) should be ≥0.1 in peripheral blood mononuclear cells
The expression level of exogenous adult hemoglobin | 18-24 Months
  Exogenous adult hemoglobin will be evaluated by globin chains and hemoglobin synthesis on peripheral blood by HPLC and the exogenous adult hemoglobin level is ≥2.0g/dL
Change from baseline in annualized frequency of packed RBC transfusions | 18-24 Months
  Compare the annualized number of pRBC transfusions before gene therapy with the Month 18 and Month 24 period after transplant, the percentage change will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Chao Liu, PHD, Principal Investigator — Shenzhen Hemogen; Sixi Liu, Professor, Principal Investigator — Shenzhen Children's Hospital
Locations (1):
- Shenzhen Children's Hospital, Shenzhen, Guangdong, China